CLINICAL TRIAL: NCT06732817
Title: Personalized Repetitive Transcranial Magnetic Stimulation for Patients with Refractory Schizophrenia: an Open-label Study
Brief Title: Personalized Dual-target RTMS for Patients with Refractory Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, MD, Anhui Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHMU-TMS-SCZ
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Schizophrenia; Transcranial Magnetic Stimulation; Functional Magnetic Resonance Imaging (fMRI)
Keywords: schizophrenia; transcranial magnetic stimulation; dual-target
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Personalized dual-target active rTMS treatment (Active Comparator): Active rTMS was sequentially administered over the left DLPFC and left TPJ sites one hour apart, for 3 weeks.
  Interventions: Device: Active rTMS was administered using a transcranial magnetic stimulator (Rapid2; MagStim).

INTERVENTIONS:
Device: Active rTMS was administered using a transcranial magnetic stimulator (Rapid2; MagStim). — Active rTMS was sequentially administered over the left DLPFC and left TPJ sites one hour apart, for 3 weeks (21 consecutive days), using a transcranial magnetic stimulator (Rapid2; MagStim) with a 70-mm air-cooled figure-of-eight coil. Stimulation at 20 Hz (2 seconds on, 28 seconds off) was applied over the left DLPFC with an intensity set at 100% of the individual resting motor threshold (RMT), delivering a total of 1,600 pulses daily. Continuous theta burst stimulation (cTBS) was applied over the left TPJ at either 100% of the individual RMT or at the highest intensity that the stimulator could deliver for this protocol (50% of maximum output). Three daily sessions of cTBS were administered, separated by two 15-minute breaks, delivering a total of 1,800 pulses daily. The coil was navigated in real-time using a frameless neuro-navigation system (Brainsight; Rogue Research, Montreal, Quebec, Canada).

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of personalized dual-target rTMS for treating patients with refractory schizophrenia and to investigate its underlying neural mechanisms using functional MRI.

The main questions it seeks to address are:

Does the dual-target rTMS protocol improve clinical symptoms in patients with refractory schizophrenia? What neural circuit changes, as assessed by functional MRI, occur following rTMS treatment?

Participants will:

Undergo personalized, dual-target rTMS treatment daily for 3 weeks. Complete baseline and post-treatment assessments, including clinical symptom scales (PANSS, HAMA, HAMD) and neuropsychological tests (MoCA, DST, VFT, Stroop Test, and AVLT).

Have structural and resting-state functional MRI scans before and after treatment.

Be monitored for any treatment-related adverse events.

DETAILED DESCRIPTION:
This open-label clinical trial aimed to evaluate the efficacy and underlying neural mechanisms of a personalized dual-target rTMS protocol for treating patients with refractory schizophrenia. Patients with refractory schizophrenia were prospectively recruited and underwent 3 weeks of rTMS treatment.

Before treatment, structural and resting-state functional MRI data were collected from each patient. Clinical symptom severity was assessed using the Positive and Negative Syndrome Scale (PANSS), Hamilton Anxiety Rating Scale (HAMA), and Hamilton Depression Rating Scale (HAMD). For patients experiencing auditory verbal hallucinations, the Auditory Hallucination Rating Scale (AHRS) was also administered. Additionally, a battery of neuropsychological tests was conducted, including the Montreal Cognitive Assessment (MoCA), Digit Span Test (DST), Verbal Fluency Test (VFT), Stroop Test, and Chinese Auditory Verbal Learning Test (AVLT).

After completing the 3-week rTMS treatment, clinical symptom severity, treatment-related adverse events, and structural and resting-state functional MRI data were reassessed.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed by independent psychiatrists using the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition;
2. disease duration longer than six years;
3. hospitalization two or more times;
4. aged 18-60 years;
5. a stable dosage of antipsychotic medication for at least four weeks before inclusion, and retention of this stable dose for the duration of the study.

Exclusion Criteria:

1. accompanied by other mental illnesses or histories;
2. pregnant;
3. a history of severe head trauma or neurological disease;
4. focal brain lesions on T1- or T2-weighted fluid-attenuated inversion-recovery MRI;
5. a history of rTMS or electroconvulsive therapy in the six months prior to the study; and
6. metal objects in the head or any other contraindication to MRI.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Positive And Negative Syndrome Scale (PANSS) | baseline and week 3 (post-treatment)
  The primary outcome was the changes in the Positive and Negative Syndrome Scale (PANSS) total scores from baseline to week 3. PANSS total score range 30 to 210, the higher scores indicate more severe symptoms.

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) subscales | baseline and week 3 (post-treatment)
  Secondary outcomes included changes in the PANSS subscales score. PANSS positive score and negative score range 7 to 49, the higher scores indicate more severe symptoms. PANSS general score range 16 to 112, the higher scores indicate more severe symptoms.
Hamilton Anxiety Rating Scale (HAMA) | baseline and week 3 (post-treatment)
  Secondary outcomes included changes in the HAMA score. HAMA scale scores range from 0 to 56 points, the higher the score indicates the more serious anxiety
Hamilton Depression Rating Scale (HAMD) | baseline and week 3 (post-treatment)
  Secondary outcomes included changes in the HAMD score. HAMA scale scores range from 0 to 50 points, the higher the score indicates the more serious depression.
Auditory Hallucination Rating Scale (AHRS) | baseline and week 3 (post-treatment)
  The changes in the Auditory Hallucination Rating Scale (AHRS) score were also included as a secondary outcome. AHRS range 0 to 41, the higher scores indicate more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No